CLINICAL TRIAL: NCT02658695
Title: Evaluation of the Relationship Between Air Bubbles Depth and Pregnancy Rate in ICSI Cycles
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Hagar Elnashar, obstetrics & gynecology resident - Ministry of health, Ain Shams Maternity Hospital
Other Study IDs: Ahmed Khairy Makled
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Good Ovarian Response; Infertility History
Keywords: ICSI; embryo transfer; air bubbles depth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: The distance between the fundal endometrial surface and air bubbles (air bubbles depth) <10 mm.
- Group 2: The distance between the fundal endometrial surface and air bubbles (air bubbles depth) >10 mm.

SUMMARY:
The aim of this work is to assess the effect of air bubbles localization inside the uterus on embryo transfer outcome in ICSI cycles.

Is there a relationship between embryo transfer outcome and the distance between fundal endometrial surface and air bubbles assessed by trans-abdominal ultrasound?

DETAILED DESCRIPTION:
All ET will be performed on day 3 after oocyte retrieval at the blastocyst stage by one operator under trans-abdominal US guidance performed by one physician, without any anesthesia or sedation with moderate bladder filling. Two embryos will be transferred using the same type of catheter which is Labotect embryo transfer catheter. It's a semirigid catheter that's less likely to induce endometrial trauma and uterine contractions.

The tip of the inner catheter will be placed approximately 1.5-2 cm from the fundal endometrial surface.The distance between the fundal endometrial surface and air bubbles will be measured and categorized as:

* Group 1: air bubbles depth <10 mm.
* Group 2: air bubbles depth >10 mm. The primary outcome will be biochemical pregnancy rate based on serum quantitative beta-hCG level at 14 days after ET. Secondary outcome will be clinical pregnancy rate using trans-vaginal US examination at 6 - 8 weeks of amenorrhea to detect the presence of fetal sac & pulsation.

ELIGIBILITY:
Inclusion Criteria:

* Women in reproductive period (age 18-38 years).
* Infertility due to bilateral tubal block or unexplained infertility programmed for ICSI.
* BMI < 25 kg/m².
* FSH level on cycle day 3 of < 12 mIU/mL

Exclusion Criteria:

* Previous failed ICSI or IVF attempts.
* Infertility due to male factors.
* Presence of an abnormal uterine cavity due to endometrial polyps, myomas distorting the uterine cavity, Mullerian malformations, endometrial synechiae, etc. (assessed by transvaginal US and/or hysterography).
* Patients with hydrosalpinx or pyosalpinx.
* Patients undergoing ET after cryopreservation.
* Patients with blood present on the catheter during the transfer procedure.
* Patients with difficult transfer or with suspicion of touching the fundus.
* Poor responders.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Eighty two women who will undergo ICSI in assisted reproductive technology unit of Ain Shams University Hospital will be enrolled in and a written informed consent will be obtained from all participants.
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
biochemical pregnancy rate | 14 days after ET
  rate of pregnant females by serum quantitative beta-hCG level at 14 days after ET

SECONDARY OUTCOMES:
clinical pregnancy rate | at 6 - 8 weeks of amenorrhea
  using trans-vaginal US examination to detect the presence of fetal sac & pulsation.

CONTACTS AND LOCATIONS:
Overall Officials: Gasser Elbishery, M.D, Study Chair — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams maternity hospital, Cairo, Egypt